CLINICAL TRIAL: NCT00300287
Title: A 56-Week Extension to a Clinical Study to Assess the Efficacy and Safety of Vildagliptin Compared to Placebo in Drug Naive Patients With Type 2 Diabetes and Mild Hyperglycemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2307E1
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; Vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

INTERVENTIONS:
Drug: Vildagliptin

SUMMARY:
This study is not being conducted in the United States. Key long-term clinical studies have shown that people with type 2 diabetes should try to achieve overall blood glucose levels as close to normal as possible. The purpose of this study is to gather data on the long-term safety and effectiveness of vildagliptin, an unapproved drug, compared to placebo in lowering overall blood glucose levels in people with type 2 diabetes who have not been previously treated with drug therapy to lower their blood sugar and whose blood glucose levels are close to normal.

ELIGIBILITY:
Inclusion Criteria:

* Completion of study CLAF237A2307 within 4 weeks of entering into the extension
* Written informed consent
* Ability to comply with all study requirements
* Blood glucose criteria must be met

Exclusion Criteria:

* Premature discontinuation from study CLAF237A2307

Min Age: 19 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2006-02-20 (Actual); Primary Completion 2007-06-26 (Actual); Study Completion 2007-06-26 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at 108 weeks

SECONDARY OUTCOMES:
Adverse event profile after 108 weeks of treatment
Change in HbA1c from week 52 to week 108
Change from baseline in fasting plasma glucose at week 108
Change in fasting plasma glucose from week 52 to week 108
Change from baseline in body weight at week 108

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Investigative Sites, Germany

REFERENCES:
- [Derived] Scherbaum WA, Schweizer A, Mari A, Nilsson PM, Lalanne G, Wang Y, Dunning BE, Foley JE. Evidence that vildagliptin attenuates deterioration of glycaemic control during 2-year treatment of patients with type 2 diabetes and mild hyperglycaemia. Diabetes Obes Metab. 2008 Nov;10(11):1114-24. doi: 10.1111/j.1463-1326.2008.00875.x. Epub 2008 Mar 18. PMID 18355325